CLINICAL TRIAL: NCT01696864
Title: Remote Rehabilitation Via the Internet in Patients After a Stroke - Physical Rehabilitation Using Biofeedback Systems to Improve Upper Extremity Function
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-12-9471-GZ-CTIL
Record Dates: First submitted 2012-09-10; First posted 2012-10-01 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2017-01

CONDITIONS: Stroke Patients

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- stroke patients - hand (Experimental): stroke patients with the ability to move their hand
  Interventions: Device: Hand tutor rehabilitation device
- stroke patient - arm (Experimental): stroke patients with the ability to move their arms
  Interventions: Device: Arm tutor rehabilitation device

INTERVENTIONS:
Device: Hand tutor rehabilitation device — A rehabilitation device for the hand
  Arms: stroke patients - hand
Device: Arm tutor rehabilitation device — A rehabilitation device for the arm
  Arms: stroke patient - arm

SUMMARY:
The objective of this study is to examine monitored rehabilitation therapy over the internet to improve upper limb function for stroke patients. Home rehabilitation for stroke patients will avoid the burden of arrival to the health facilities, making it easier on them and improve their quality of life and the lives of their caregivers. To achieve this goal the investigators will examine the effectiveness and feasibility of home rehabilitation system of upper limb, consisting of ergonomic accessories (hand and arm tutors).

The quantitative indices will be based on the quantitative clinical measures that are used in regular evaluations of stroke patients and function and range of motion indices as received from the system.

ELIGIBILITY:
Inclusion Criteria:

* Stroke patients who had at least eight conventional rehabilitation treatments lasted at least until a month before the start of the experiment,
* not affected cognitively (to be determined by the score on the mini mental exam greater than 23).
* patients have daily access to a computer and the Internet, and use a personal caregiver or family member can supervise the use of the system.

Exclusion Criteria:

* Global or sensory aphasia, unilateral spatial neglect, apraxia and other acute neurological or orthopedic conditions.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-03; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment upper extremity part (FMA) | 10 minutes
  The FMA assesses the motor impairment of the upper extremity after stroke. Each movement is graded on a 3-point scale, and the total score for the upper extremity ranges from 0-60 points where a higher score represents more active movements. An additional part assesses the coordination of the affected upper extremity and the score ranges between 0-6 where a higher score represents poorer coordination ability. This test is one of the most commonly used instruments in rehabilitation and its validity and reliability have been well established
Arm and Hand Activity Inventory (CAHAI) | 10 minutes
  The test assesses the functional ability of the affected arm and hand of people with stroke. The abbreviated version includes 7 functional activities (e.g. open a jar of coffee) that require bilateral use of the upper extremities as well various types of grip. The score range between1 and 7
Motor Activity Log (MAL) | 10 minutes
  The MAL consist of a semi structured interview for the patient to assess the use of the paretic arm and hand during daily activities. Two scores on a scale of 1 -5, are given for each activity;for the amount of use (AOU) and for the quality of movement (QOM). Usability of the system i.e. ease of use of the system
System Usability Scale (SUS) | 10 minutes
  This questionnaire includes 10 items rated on a 5 points scale, which provide a global view of subjective assessment of a system's usability. The item scores were calculated to give an overall score ranging from 10 to 100 points. The SUS has been shown to be a robust and reliable evaluation tool
Box& Block Test of Manual Dexterity | 10 minutes
  This is a valid and reliable test which is used to assess hand dexterity. In addition it is used to assess endurance of the upper extremity. The subject is asked to transfer cubes, above a partition, from one side of a box to the other for one minute with both hands. The score is the number of cubes that were transferred. In addition: Range of motion of fingers, wrist elbow and shoulder as measured by the devices

CONTACTS AND LOCATIONS:
Overall Officials: Gabi Zeilig, Dr., Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center rehabilitation facility, Ramat Gan, Israel